CLINICAL TRIAL: NCT00463606
Title: A 12-week, Multicenter, Randomized, Double-Blind, Parallel-Group Study of the Combination of ABT-335 and Rosuvastatin Compared to ABT-335 and Rosuvastatin Monotherapy in Subjects With Type IIa and IIb Dyslipidemia
Brief Title: A Multicenter Study Comparing the Safety and Efficacy of ABT-335 and Rosuvastatin Calcium Combination Therapy to Monotherapy in Subjects With Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M06-844
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Hypercholesterolemia; Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium; fenofibric acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABT-335 and Rosuvastatin Calcium (Experimental): ABT-335 135mg in combination with rosuvastatin calcium 5mg administered orally, once daily for 12 weeks
  Interventions: Drug: ABT-335 and rosuvastatin calcium
- ABT-335 (Active Comparator): ABT-335 135mg monotherapy administered orally, once daily for 12 weeks
  Interventions: Drug: ABT-335
- Rosuvastatin Calcium (Active Comparator): Rosuvastatin calcium 5mg monotherapy administered orally, once daily for 12 weeks
  Interventions: Drug: rosuvastatin calcium

INTERVENTIONS:
Drug: ABT-335 and rosuvastatin calcium — ABT-335 135 mg in combination with rosuvastatin calcium 5 mg administered orally, once daily for 12 weeks
  Other Names: ABT-335 / Rosuvastatin Combination (ABT-143)
  Arms: ABT-335 and Rosuvastatin Calcium
Drug: ABT-335 — ABT-335 135 mg monotherapy administered orally, once daily for 12 weeks
  Other Names: fenofibric acid
  Arms: ABT-335
Drug: rosuvastatin calcium — Rosuvastatin calcium 5 mg monotherapy administered orally, once daily for 12 weeks
  Other Names: Rosuvastatin
  Arms: Rosuvastatin Calcium

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ABT-335 and rosuvastatin calcium combination therapy to monotherapy in subjects with dyslipidemia.

DETAILED DESCRIPTION:
There are 3 treatment groups in the study: ABT-335 135 mg in combination with rosuvastatin 5 mg, ABT-335 135 mg monotherapy, and rosuvastatin 5 mg monotherapy. The 3 primary outcome measures only compare 2 of the treatment groups for each variable (mean percent change in HDL-C and TG comparing ABT-335 135 mg in combination with rosuvastatin 5 mg to rosuvastatin 5 mg monotherapy, and mean percent change in LDL-C comparing ABT-335 135 mg in combination with rosuvastatin 5 mg to ABT-335 135 mg monotherapy. The 6 secondary outcome measures only compare 2 of the treatment groups for each variable (mean percent change in Non-HDL-C comparing ABT-335 135 mg in combination with rosuvastatin 5 mg to ABT-335 135 mg monotherapy, mean percent change in Non-HDL-C, VLDL-C, ApoB, and Total Cholesterol comparing ABT-335 135 mg in combination with rosuvastatin 5 mg to rosuvastatin 5 mg monotherapy, and median percent change in hsCRP comparing ABT-335 135 mg in combination with rosuvastatin 5 mg to rosuvastatin 5 mg monotherapy).

ELIGIBILITY:
Inclusion Criteria

* Adult male and female participants who voluntarily sign the informed consent.
* Fasting lipid results following greater than 12-hour fasting period:

  * Triglycerides level greater than or equal to 150 mg/dL,
  * High-density lipoprotein cholesterol less than 40 mg/dL for males and less than 50 mg/dL for females, and
  * Low-density lipoprotein cholesterol greater than or equal to 130 mg/dL.
* Participant must agree to utilize adequate birth control methods and adhere to the American Heart Association (AHA) diet.

Exclusion Criteria

* Participants with unstable medical conditions, medical conditions considered inappropriate in a clinical trial, or participants who are taking excluded concomitant medications are not allowed in the study.
* Participants receiving coumarin anticoagulants or systemic cyclosporine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (168):
- United States (168):
  - Site Reference ID/Investigator# 5469, Birmingham, Alabama
  - Site Reference ID/Investigator# 4428, Birmingham, Alabama
  - Site Reference ID/Investigator# 4985, Birmingham, Alabama
  - Site Reference ID/Investigator# 4493, Huntsville, Alabama
  - Site Reference ID/Investigator# 4510, Huntsville, Alabama
  - Site Reference ID/Investigator# 4431, Ozark, Alabama
  - Site Reference ID/Investigator# 4519, Tuscaloosa, Alabama
  - Site Reference ID/Investigator# 4395, Chandler, Arizona
  - Site Reference ID/Investigator# 4483, Gilbert, Arizona
  - Site Reference ID/Investigator# 4411, Scottsdale, Arizona
  - Site Reference ID/Investigator# 4417, Little Rock, Arkansas
  - Site Reference ID/Investigator# 4702, Anaheim, California
  - Site Reference ID/Investigator# 5593, Chula Vista, California
  - Site Reference ID/Investigator# 4503, Concord, California
  - Site Reference ID/Investigator# 4530, Encinitas, California
  - Site Reference ID/Investigator# 4458, Fair Oaks, California
  - Site Reference ID/Investigator# 4542, Fresno, California
  - Site Reference ID/Investigator# 4574, Fresno, California
  - Site Reference ID/Investigator# 4441, Lincoln, California
  - Site Reference ID/Investigator# 4432, Long Beach, California
  - Site Reference ID/Investigator# 5579, Los Angeles, California
  - Site Reference ID/Investigator# 4980, Norwalk, California
  - Site Reference ID/Investigator# 4392, Sacramento, California
  - Site Reference ID/Investigator# 4896, Sacramento, California
  - Site Reference ID/Investigator# 5582, San Diego, California
  - Site Reference ID/Investigator# 6236, West Hills, California
  - Site Reference ID/Investigator# 4442, Aurora, Colorado
  - Site Reference ID/Investigator# 4419, Colorado Springs, Colorado
  - Site Reference ID/Investigator# 4391, Waterbury, Connecticut
  - Site Reference ID/Investigator# 4401, Coral Gables, Florida
  - Site Reference ID/Investigator# 4453, Fort Lauderdale, Florida
  - Site Reference ID/Investigator# 4490, Holly Hill, Florida
  - Site Reference ID/Investigator# 4420, Hollywood, Florida
  - Site Reference ID/Investigator# 5011, Jacksonville, Florida
  - Site Reference ID/Investigator# 4444, Jacksonville, Florida
  - Site Reference ID/Investigator# 4399, Jupiter, Florida
  - Site Reference ID/Investigator# 4433, Kissimmee, Florida
  - Site Reference ID/Investigator# 4469, Largo, Florida
  - Site Reference ID/Investigator# 4525, Melbourne, Florida
  - Site Reference ID/Investigator# 4477, Miami, Florida
  - Site Reference ID/Investigator# 4430, New Port Richey, Florida
  - Site Reference ID/Investigator# 4409, New Smyrna Beach, Florida
  - Site Reference ID/Investigator# 4416, Ocala, Florida
  - Site Reference ID/Investigator# 4528, Ocala, Florida
  - Site Reference ID/Investigator# 5103, Orlando, Florida
  - Site Reference ID/Investigator# 4446, Ormond Beach, Florida
  - Site Reference ID/Investigator# 4524, Pensacola, Florida
  - Site Reference ID/Investigator# 4505, Sarasota, Florida
  - Site Reference ID/Investigator# 5580, Sarasota, Florida
  - Site Reference ID/Investigator# 4494, West Palm Beach, Florida
  - Site Reference ID/Investigator# 4407, West Palm Beach, Florida
  - Site Reference ID/Investigator# 4512, Winter Haven, Florida
  - Site Reference ID/Investigator# 5478, Blue Ridge, Georgia
  - Site Reference ID/Investigator# 4388, Decatur, Georgia
  - Site Reference ID/Investigator# 4511, Dunwoody, Georgia
  - Site Reference ID/Investigator# 4981, Roswell, Georgia
  - Site Reference ID/Investigator# 4448, Roswell, Georgia
  - Site Reference ID/Investigator# 4497, Suwanee, Georgia
  - Site Reference ID/Investigator# 4439, Woodstock, Georgia
  - Site Reference ID/Investigator# 4472, Arlington Heights, Illinois
  - Site Reference ID/Investigator# 5585, Chicago, Illinois
  - Site Reference ID/Investigator# 4520, Peoria, Illinois
  - Site Reference ID/Investigator# 4527, Avon, Indiana
  - Site Reference ID/Investigator# 4485, Evansville, Indiana
  - Site Reference ID/Investigator# 4445, Indianapolis, Indiana
  - Site Reference ID/Investigator# 4438, Lafayette, Indiana
  - Site Reference ID/Investigator# 5010, Newburgh, Indiana
  - Site Reference ID/Investigator# 4403, Iowa City, Iowa
  - Site Reference ID/Investigator# 4393, Arkansas City, Kansas
  - Site Reference ID/Investigator# 4526, Overland Park, Kansas
  - Site Reference ID/Investigator# 4423, Wichita, Kansas
  - Site Reference ID/Investigator# 4424, Wichita, Kansas
  - Site Reference ID/Investigator# 5027, Lexington, Kentucky
  - Site Reference ID/Investigator# 4471, Louisville, Kentucky
  - Site Reference ID/Investigator# 4406, New Orleans, Louisiana
  - Site Reference ID/Investigator# 4509, Slidell, Louisiana
  - Site Reference ID/Investigator# 5635, Auburn, Maine
  - Site Reference ID/Investigator# 4502, Scarborough, Maine
  - Site Reference ID/Investigator# 5070, Baltimore, Maryland
  - Site Reference ID/Investigator# 4412, Haverhill, Massachusetts
  - Site Reference ID/Investigator# 4487, Springfield, Massachusetts
  - Site Reference ID/Investigator# 5533, Ann Arbor, Michigan
  - Site Reference ID/Investigator# 6237, Ann Arbor, Michigan
  - Site Reference ID/Investigator# 5583, Portage, Michigan
  - Site Reference ID/Investigator# 4480, Brooklyn Center, Minnesota
  - Site Reference ID/Investigator# 4515, Jackson, Mississippi
  - Site Reference ID/Investigator# 4492, Olive Branch, Mississippi
  - Site Reference ID/Investigator# 5636, Tupelo, Mississippi
  - Site Reference ID/Investigator# 4499, City of Saint Peters, Missouri
  - Site Reference ID/Investigator# 4500, Kansas City, Missouri
  - Site Reference ID/Investigator# 4979, Billings, Montana
  - Site Reference ID/Investigator# 4481, Missoula, Montana
  - Site Reference ID/Investigator# 4460, Las Vegas, Nevada
  - Site Reference ID/Investigator# 4466, Las Vegas, Nevada
  - Site Reference ID/Investigator# 5484, Las Vegas, Nevada
  - Site Reference ID/Investigator# 5444, Concord, New Hampshire
  - Site Reference ID/Investigator# 4908, Elizabeth, New Jersey
  - Site Reference ID/Investigator# 4504, South Bound Brook, New Jersey
  - Site Reference ID/Investigator# 4394, Toms River, New Jersey
  - Site Reference ID/Investigator# 4402, Trenton, New Jersey
  - Site Reference ID/Investigator# 4427, Albuquerque, New Mexico
  - Site Reference ID/Investigator# 4463, Bronxville, New York
  - Site Reference ID/Investigator# 4415, New York, New York
  - Site Reference ID/Investigator# 4440, Rochester, New York
  - Site Reference ID/Investigator# 4464, Syracuse, New York
  - Site Reference ID/Investigator# 4425, Williamsville, New York
  - Site Reference ID/Investigator# 4473, Asheville, North Carolina
  - Site Reference ID/Investigator# 4531, Charlotte, North Carolina
  - Site Reference ID/Investigator# 4396, Charlotte, North Carolina
  - Site Reference ID/Investigator# 5494, Hickory, North Carolina
  - Site Reference ID/Investigator# 4479, Morehead City, North Carolina
  - Site Reference ID/Investigator# 4461, Raleigh, North Carolina
  - Site Reference ID/Investigator# 4498, Salisbury, North Carolina
  - Site Reference ID/Investigator# 4405, Statesville, North Carolina
  - Site Reference ID/Investigator# 4476, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 4390, Cincinnati, Ohio
  - Site Reference ID/Investigator# 4400, Cincinnati, Ohio
  - Site Reference ID/Investigator# 4501, Cincinnati, Ohio
  - Site Reference ID/Investigator# 4517, Cincinnati, Ohio
  - Site Reference ID/Investigator# 5584, Columbus, Ohio
  - Site Reference ID/Investigator# 4410, Mogadore, Ohio
  - Site Reference ID/Investigator# 4443, Sandusky, Ohio
  - Site Reference ID/Investigator# 4523, Warren, Ohio
  - Site Reference ID/Investigator# 4488, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 4451, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 4422, Tulsa, Oklahoma
  - Site Reference ID/Investigator# 4482, Tulsa, Oklahoma
  - Site Reference ID/Investigator# 4467, Medford, Oregon
  - Site Reference ID/Investigator# 4470, Carlisle, Pennsylvania
  - Site Reference ID/Investigator# 5581, Downingtown, Pennsylvania
  - Site Reference ID/Investigator# 4434, Feasterville, Pennsylvania
  - Site Reference ID/Investigator# 4478, Harleysville, Pennsylvania
  - Site Reference ID/Investigator# 4436, Jersey Shore, Pennsylvania
  - Site Reference ID/Investigator# 4397, Lansdale, Pennsylvania
  - Site Reference ID/Investigator# 4426, Melrose Park, Pennsylvania
  - Site Reference ID/Investigator# 4894, Newtown, Pennsylvania
  - Site Reference ID/Investigator# 4496, Penndel, Pennsylvania
  - Site Reference ID/Investigator# 4404, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 4437, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 4387, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 4447, Warminster, Pennsylvania
  - Site Reference ID/Investigator# 4506, Charleston, South Carolina
  - Site Reference ID/Investigator# 5443, Greenville, South Carolina
  - Site Reference ID/Investigator# 4484, Greer, South Carolina
  - Site Reference ID/Investigator# 4455, Moncks Corner, South Carolina
  - Site Reference ID/Investigator# 4513, Mt. Pleasant, South Carolina
  - Site Reference ID/Investigator# 4521, Simpsonville, South Carolina
  - Site Reference ID/Investigator# 4982, Summerville, South Carolina
  - Site Reference ID/Investigator# 5586, Sioux Falls, South Dakota
  - Site Reference ID/Investigator# 4435, Jackson, Tennessee
  - Site Reference ID/Investigator# 4454, Johnson City, Tennessee
  - Site Reference ID/Investigator# 4529, Nashville, Tennessee
  - Site Reference ID/Investigator# 5454, Arlington, Texas
  - Site Reference ID/Investigator# 5578, Houston, Texas
  - Site Reference ID/Investigator# 5669, Houston, Texas
  - Site Reference ID/Investigator# 4893, San Antonio, Texas
  - Site Reference ID/Investigator# 4429, San Antonio, Texas
  - Site Reference ID/Investigator# 4457, San Antonio, Texas
  - Site Reference ID/Investigator# 4465, San Antonio, Texas
  - Site Reference ID/Investigator# 4508, San Antonio, Texas
  - Site Reference ID/Investigator# 4892, San Antonio, Texas
  - Site Reference ID/Investigator# 5948, San Antonio, Texas
  - Site Reference ID/Investigator# 4413, Temple, Texas
  - Site Reference ID/Investigator# 4456, Falls Church, Virginia
  - Site Reference ID/Investigator# 4459, Richmond, Virginia
  - Site Reference ID/Investigator# 4408, Richmond, Virginia
  - Site Reference ID/Investigator# 4421, Lakewood, Washington
  - Site Reference ID/Investigator# 4468, Madison, Wisconsin

REFERENCES:
- [Derived] Rosenson RS, Carlson DM, Kelly MT, Setze CM, Hirshberg B, Stolzenbach JC, Williams LA. Achievement of lipid targets with the combination of rosuvastatin and fenofibric Acid in patients with type 2 diabetes mellitus. Cardiovasc Drugs Ther. 2011 Feb;25(1):47-57. doi: 10.1007/s10557-010-6273-5. PMID 21174145
- [Derived] Roth EM, Rosenson RS, Carlson DM, Fukumoto SM, Setze CM, Blasetto JW, Khurmi NS, Stolzenbach JC, Williams LA. Efficacy and safety of rosuvastatin 5 mg in combination with fenofibric acid 135 mg in patients with mixed dyslipidemia - a phase 3 study. Cardiovasc Drugs Ther. 2010 Dec;24(5-6):421-8. doi: 10.1007/s10557-010-6266-4. PMID 20953684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 760 participants were randomized at 144 sites in the United States, and 758 participants were treated between 07 June 2007 and 10 February 2008. Two participants were randomized but not treated: 1 was lost to follow-up and 1 was withdrawn at the investigator's discretion.
Pre-assignment Details: A total of 168 study sites screened participants, wtih 144 of these sites randomizing participants.
Period: Overall Study
Arm/Group | ABT-335 and Rosuvastatin Calcium | ABT-335 | Rosuvastatin Calcium
Started | 253 | 254 | 251
Completed | 212 | 220 | 231
Not Completed | 41 | 34 | 20
Not completed — Adverse Event | 21 | 18 | 11
Not completed — Withdrawal by Subject | 11 | 11 | 5
Not completed — Lost to Follow-up | 2 | 2 | 3
Not completed — Subject noncompliance | 1 | 1 | 0
Not completed — Subject moved out of town | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Sponsor request | 0 | 1 | 0
Not completed — Exclusion criteria violation | 2 | 0 | 0
Not completed — Coordinator error | 1 | 0 | 0
Not completed — Patient randomized in error | 1 | 0 | 0
Not completed — Participation in another ABT-335 trial | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 and Rosuvastatin Calcium | ABT-335 | Rosuvastatin Calcium | Total
Number analyzed (Participants) | 253 | 254 | 251 | 758
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 194 | 203 | 205 | 602
  >=65 years | 59 | 51 | 46 | 156
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.30) | 54.4 (11.24) | 55.3 (10.71) | 55.3 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 144 | 150 | 455
  Male | 92 | 110 | 101 | 303
Region of Enrollment [Number; unit: participants]
  United States | 253 | 254 | 251 | 758

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline to the Final Visit in High-density Lipoprotein Cholesterol (HDL-C) (Full Analysis Set)
Description: The mean percent change from baseline to the final visit in High-density lipoprotein cholesterol (HDL-C), with ABT-335 135 mg in combination with rosuvastatin 5 mg versus rosuvastatin 5 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline and at least 1 post-baseline value for high-density lipoprotein cholesterol. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | Rosuvastatin Calcium
Number analyzed (Participants) | 236 | 241
percent change | 23.0 (1.33) | 12.4 (1.32)

2. Primary Outcome: Mean Percent Change From Baseline to the Final Visit in Triglycerides (Full Analysis Set)
Description: The mean percent change from baseline to the final visit in triglycerides, with ABT-335 135 mg in combination with rosuvastatin 5 mg versus rosuvastatin 5 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for triglycerides. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | Rosuvastatin Calcium
Number analyzed (Participants) | 236 | 241
percent change | -40.3 (1.89) | -17.5 (1.88)

3. Primary Outcome: Mean Percent Change From Baseline to the Final Visit in Low-density Lipoprotein Cholesterol (LDL-C) (Full Analysis Set)
Description: The mean percent change from baseline to the final visit in low-density lipoprotein cholesterol (LDL-C), with ABT-335 135 mg in combination with rosuvastatin 5 mg versus ABT-335 135 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for low-density lipoprotein cholesterol. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | ABT-335
Number analyzed (Participants) | 236 | 245
percent change | -28.7 (1.33) | -4.1 (1.31)

4. Secondary Outcome: Mean Percent Change From Baseline to the Final Visit in Non-high-density Lipoprotein Cholesterol (Non-HDL-C), With ABT-335 135 mg in Combination With Rosuvastatin 5 mg Versus ABT-335 135 mg Monotherapy (Full Analysis Set)
Description: The mean percent change from baseline to the final visit in non-high-density lipoprotein cholesterol (non-HDL-C), with ABT-335 135 mg in combination with rosuvastatin 5 mg versus ABT-335 135 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for non-HDL-C. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | ABT-335
Number analyzed (Participants) | 236 | 245
percent change | -37.4 (1.06) | -16.0 (1.05)

5. Secondary Outcome: Mean Percent Change From Baseline to the Final Visit in Non-high-density Lipoprotein Cholesterol (Non-HDL-C), With ABT-335 135 mg in Combination With Rosuvastatin 5 mg Versus Rosuvastatin 5 mg Monotherapy (Full Analysis Set)
Description: The mean percent change from baseline to the final visit in non-high-density lipoprotein cholesterol (non-HDL-C), with ABT-335 135 mg in combination with rosuvastatin 5 mg versus rosuvastatin 5 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | Rosuvastatin Calcium
Number analyzed (Participants) | 236 | 241
percent change | -37.4 (1.06) | -31.8 (1.05)

6. Secondary Outcome: Mean Percent Change From Baseline to the Final Visit in Very-low-density Lipoprotein Cholesterol (VLDL-C) (Full Analysis Set)
Description: The mean percent change from baseline to the final visit in very-low-density lipoprotein cholesterol (VLDL-C), with ABT-335 135 mg in combination with rosuvastatin 5 mg versus rosuvastatin 5 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for VLDL-C. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | Rosuvastatin Calcium
Number analyzed (Participants) | 235 | 239
percent change | -41.3 (3.56) | -22.2 (3.53)

7. Secondary Outcome: Mean Percent Change From Baseline to the Final Visit in Apolipoprotein B (ApoB) (Full Analysis Set)
Description: The mean percent change from baseline to the final visit in apolipoprotein B (ApoB), with ABT-335 135 mg in combination with rosuvastatin 5 mg versus rosuvastatin 5 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for ApoB. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | Rosuvastatin Calcium
Number analyzed (Participants) | 233 | 238
percent change | -30.9 (1.00) | -26.4 (0.99)

8. Secondary Outcome: Median Percent Change From Baseline to the Final Visit in High Sensitivity C-reactive Protein (hsCRP) (Full Analysis Set)
Description: The median percent change from baseline to the final visit in high sensitivity C-reactive protein (hsCRP), with ABT-335 135 mg in combination with rosuvastatin 5 mg versus rosuvastatin 5 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for hsCRP. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | Rosuvastatin Calcium
Number analyzed (Participants) | 235 | 240
percent change | -28.0 [-49.1 to 9.0] | -11.4 [-37.4 to 26.8]

9. Secondary Outcome: Mean Percent Change From Baseline to the Final Visit in Total Cholesterol (Full Analysis Set)
Description: The mean percent change from baseline to the final visit in total cholesterol, with ABT-335 135 mg in combination with rosuvastatin 5 mg versus rosuvastatin 5 mg monotherapy.
Time Frame: Baseline to 12 Weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 post-baseline value for total cholesterol. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 and Rosuvastatin Calcium | Rosuvastatin Calcium
Number analyzed (Participants) | 236 | 241
percent change | -28.1 (0.85) | -25.0 (0.84)

ADVERSE EVENTS:
Time Frame: Up to 23 weeks
Description: All adverse events reported from the time of study drug administration until 30 days following discontinuation of study drug were collected. Serious adverse events were collected from the time the participant signed the informed consent until 30 days following discontinuation of study drug.
Arm/Group | ABT-335 and Rosuvastatin Calcium | ABT-335 | Rosuvastatin Calcium
Serious Adverse Events (participants affected / at risk) | 7/253 | 6/254 | 4/251
Other Adverse Events (participants affected / at risk) | 52/253 | 41/254 | 45/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 and Rosuvastatin Calcium (N=253) | ABT-335 (N=254) | Rosuvastatin Calcium (N=251)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Cyst (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 and Rosuvastatin Calcium (N=253) | ABT-335 (N=254) | Rosuvastatin Calcium (N=251)
Dyspepsia (Gastrointestinal disorders) | 16 | 6 | 2
Nasopharyngitis (Infections and infestations) | 6 | 15 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 11 | 14
Headache (Nervous system disorders) | 28 | 23 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.